CLINICAL TRIAL: NCT04453332
Title: Effects of Oral and Non-oral Hormonal Therapy on Cardiovascular Risk and Body Composition Parameters in Postmenopausal Women
Brief Title: Effects of Hormone Replacement Therapy on Cardiovascular Risk and Body Composition Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0363
Record Dates: First submitted 2020-06-23; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Menopause; Hormone Replacement Therapy
Keywords: Menopause; Hormone therapy; Body composition; Metabolism
MeSH Terms: interventions — Estradiol

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral hormone therapy (Active Comparator): Estradiol 1mg and micronized natural progesterone 200mg 14 days a month (oral)
  Interventions: Drug: Oral hormone therapy (estradiol and micronized natural progesterone)
- Non-oral hormone therapy (Active Comparator): Percutaneous estradiol gel 1.5mg and micronized progesterone 200mg vaginal 14 days a month (non-oral)
  Interventions: Drug: Non-oral hormone therapy (estradiol and micronized natural progesterone)

INTERVENTIONS:
Drug: Oral hormone therapy (estradiol and micronized natural progesterone) — Oral hormone therapy - estradiol 1mg every day and micronized natural progesterone 200mg only 14 days a month
  Arms: Oral hormone therapy
Drug: Non-oral hormone therapy (estradiol and micronized natural progesterone) — Percutaneous estradiol gel 1.5mg every day and micronized progesterone 200mg vaginal only 14 days a month
  Arms: Non-oral hormone therapy

SUMMARY:
Menopause is defined as the last episode of menstrual bleeding, resulting from the interruption of ovarian function by follicular depletion. It is characterized by the presence of amenorrhea associated with increased levels of FSH and low levels of estradiol. The decline in estrogenic levels is associated with several organic changes, from vasomotor symptoms to impaired bone mass and urogenital atrophy. Although for some patients menopause is asymptomatic or oligosymptomatic, many women experience intense symptoms, which profoundly affect quality of life.

Proper assessment and treatment of postmenopausal women can significantly improve climacteric symptoms. Target tissue, hormone therapy regimen and variations between patients will influence the effects of treatment. Regarding estrogen, the main factors that influence the therapeutic response are the type of hormone used, the dose and the route of administration. The skin metabolizes only a small part of estradiol. Thus, the transdermal route reaches adequate therapeutic levels from a lower dose of estrogen.

The present study aims to evaluate and compare the effects of low dose of oral estradiol associated with oral progesterone and transdermal estradiol associated with vaginal progesterone on variables related to inflammation, coagulation and body composition parameters.

DETAILED DESCRIPTION:
Hormone therapy (HT) was available since 1942 in tablets containing conjugated equine estrogens. Since the 1970s, it has been recommended to add progestogens to the treatment of women with a uterus to prevent endometrial hyperplasia. HT has been shown to be very effective in climacteric syndrome, relieving 90% of hot flushes that affect women in the menopausal transition.

Target tissue, HT regimen and variations between patients will influence the effects of treatment. Regarding estrogen, the main factors that influence the therapeutic response are the type of hormone used, the dose and the route of administration. The most physiological type of estrogen is 17β estradiol, available in the form of gel and adhesive. The skin metabolizes only a small part of estradiol. Thus, the transdermal route reaches adequate therapeutic levels from a lower dose of estrogen. Also, the transdermal route prevents the first hepatic passage, resulting in more stable levels of estradiol in the circulation, without supraphysiological liver concentrations. The bioavailability of estrogen after undergoing metabolism in the liver is approximately 2 to 10% of the total administered. This hepatic passage can result in greater variability in hormone levels, as well as activation of prothrombotic and inflammatory factors. In addition, hepatic metabolism can change the therapeutic effects of estrogen and other pharmacological agents.

The present study aims to evaluate and compare the effects of low dose of oral estradiol associated with oral progesterone and transdermal estradiol associated with vaginal progesterone on variables related to inflammation, coagulation and body composition parameters. This is a prospective randomized controlled study, and the study population includes postmenopausal patients with climacteric symptoms, who have not been using hormone therapy for at least three months. Patients will receive three months of oral hormonal treatment (estradiol 1mg and micronized natural progesterone 200mg 14 days a month) and three months of non-oral hormonal treatment (percutaneous estradiol gel 1.5mg and micronized progesterone 200mg vaginal 14 days a month).

Patients with climacteric symptoms who meet the inclusion and the exclusion criteria will be included in the study. The entire sample will receive both hormonal therapies sequentially and the patients will be divided between the groups (oral therapy and non-oral therapy) to start the study by random allocation. There will be no period of suspension between treatments, that is, at the end of the first three months of the study, the group initially treated with oral therapy starts receiving non-oral treatment for another three months, and the group initially treated with non-oral therapy starts to receive oral therapy also for another three months.

This project has already been approved by the Research Ethics Committee of the Hospital de Clínicas de Porto Alegre. Post-informed written consent will be obtained from all patients, in accordance with health research standards.

The results will be presented as means and standard deviation or medians and interquartile range. Analysis of variance for latin square will be used to evaluate carryover effect. Two-way ANOVA for repeated samples will be used to compare baseline conditions and the two treatments. Bonferroni's adjustment will be used for multiple comparisons. Bivariate correlations between continuous numerical variables will be examined using Pearson or Spearman correlation coefficients, according to the Gaussian or non-Gaussian nature of the variable, respectively. Statistical analysis will be performed using Statistical Package for Social Sciences (SPSS, Chicago, IL, USA), with a value of p <0.05 being considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Six months or more of amenorrhea and FSH levels> or = at 35 mIU / ml;
* Menopause for a maximum of three years;
* Mammography and cytology of recent cervix (from the last 12 months);
* Signature of the Informed Consent Form.

Exclusion Criteria:

* Menopause age below 40 years;
* Use of hormonal therapy in the three months preceding the study;
* Uncontrolled diabetes mellitus;
* Endometrial thickening (endometrial thickness greater than 0.5 cm);
* Neoplasm of breast, colon or endometrium;
* History of thromboembolism or established cardiovascular disease;
* Previous hysterectomy;
* Active smoking;
* Use of medication to treat osteoporosis in the last 12 months: bisphosphonates, denosumab, teriparatide, SERMs (selective estrogen receptor agonist).

Ages: 40 Years to 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2015-10-09 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in body composition parameters | Before hormone therapy and after 3 and 6 months of treatment
  Lean mass (kilograms) evaluated by dual energy X-ray absorptiometry (DXA)
Change in body composition parameters | Before hormone therapy and after 3 and 6 months of treatment
  Fat mass (kilograms) evaluated by dual energy X-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Lipid profile | Before hormone therapy and after 3 and 6 months of treatment
  HDL, LDL, triglycerides (evaluated by blood sample)
Serum glucose | Before hormone therapy and after 3 and 6 months of treatment
  (evaluated by blood sample)
Blood pressure | Before hormone therapy and after 3 and 6 months of treatment
Weight | Before hormone therapy and after 3 and 6 months of treatment
  With body mass index (kg/m²)
Physical activity | Before hormone therapy and after 3 and 6 months of treatment
  Evaluated by pedometer
Bone mineral density (g/cm²) | Before hormone therapy and after 3 and 6 months of treatment
  Evaluated by dual energy X-ray absorptiometry (DXA)
Bone metabolism | Before hormone therapy
  Calcium, phosphorus, PTH, albumin, 25 OH vitamin D (evaluated by blood sample)

CONTACTS AND LOCATIONS:
Overall Officials: Poli Mara Spritzer, PhD, Principal Investigator — Federal University of Rio Grande do Sul, Porto Alegre, Brazil
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] LaCroix AZ, Chlebowski RT, Manson JE, Aragaki AK, Johnson KC, Martin L, Margolis KL, Stefanick ML, Brzyski R, Curb JD, Howard BV, Lewis CE, Wactawski-Wende J; WHI Investigators. Health outcomes after stopping conjugated equine estrogens among postmenopausal women with prior hysterectomy: a randomized controlled trial. JAMA. 2011 Apr 6;305(13):1305-14. doi: 10.1001/jama.2011.382. PMID 21467283
- [Background] L'hermite M, Simoncini T, Fuller S, Genazzani AR. Could transdermal estradiol + progesterone be a safer postmenopausal HRT? A review. Maturitas. 2008 Jul-Aug;60(3-4):185-201. doi: 10.1016/j.maturitas.2008.07.007. Epub 2008 Sep 5. PMID 18775609
- [Background] Rovinski D, Ramos RB, Fighera TM, Casanova GK, Spritzer PM. Risk of venous thromboembolism events in postmenopausal women using oral versus non-oral hormone therapy: A systematic review and meta-analysis. Thromb Res. 2018 Aug;168:83-95. doi: 10.1016/j.thromres.2018.06.014. Epub 2018 Jun 19. PMID 29936403
- [Background] Modena MG, Sismondi P, Mueck AO, Kuttenn F, Lignieres Bd, Verhaeghe J, Foidart JM, Caufriez A, Genazzani AR; TREAT. New evidence regarding hormone replacement therapies is urgently required transdermal postmenopausal hormone therapy differs from oral hormone therapy in risks and benefits. Maturitas. 2005 Sep 16;52(1):1-10. doi: 10.1016/j.maturitas.2005.05.003. PMID 15963666
- [Background] Casanova G, Radavelli S, Lhullier F, Spritzer PM. Effects of nonoral estradiol-micronized progesterone or low-dose oral estradiol-drospirenone therapy on metabolic variables and markers of endothelial function in early postmenopause. Fertil Steril. 2009 Aug;92(2):605-12. doi: 10.1016/j.fertnstert.2008.06.049. Epub 2008 Aug 15. PMID 18706557
- [Background] Casanova G, Spritzer PM. Effects of micronized progesterone added to non-oral estradiol on lipids and cardiovascular risk factors in early postmenopause: a clinical trial. Lipids Health Dis. 2012 Oct 9;11:133. doi: 10.1186/1476-511X-11-133. PMID 23046709
- [Background] Lara S, Casanova G, Spritzer PM. Influence of habitual physical activity on body composition, fat distribution and metabolic variables in early postmenopausal women receiving hormonal therapy. Eur J Obstet Gynecol Reprod Biol. 2010 May;150(1):52-6. doi: 10.1016/j.ejogrb.2010.02.007. Epub 2010 Feb 26. PMID 20189290
- [Background] Casanova G, Bossardi Ramos R, Ziegelmann P, Spritzer PM. Effects of low-dose versus placebo or conventional-dose postmenopausal hormone therapy on variables related to cardiovascular risk: a systematic review and meta-analyses of randomized clinical trials. J Clin Endocrinol Metab. 2015 Mar;100(3):1028-37. doi: 10.1210/jc.2014-3301. Epub 2014 Dec 16. PMID 25514104
- [Background] Goodman MP. Are all estrogens created equal? A review of oral vs. transdermal therapy. J Womens Health (Larchmt). 2012 Feb;21(2):161-9. doi: 10.1089/jwh.2011.2839. Epub 2011 Oct 19. PMID 22011208
- [Background] Rossouw JE, Anderson GL, Prentice RL, LaCroix AZ, Kooperberg C, Stefanick ML, Jackson RD, Beresford SA, Howard BV, Johnson KC, Kotchen JM, Ockene J; Writing Group for the Women's Health Initiative Investigators. Risks and benefits of estrogen plus progestin in healthy postmenopausal women: principal results From the Women's Health Initiative randomized controlled trial. JAMA. 2002 Jul 17;288(3):321-33. doi: 10.1001/jama.288.3.321. PMID 12117397